CLINICAL TRIAL: NCT03452007
Title: Functional Mapping With Lumbosacral Epidural Stimulation for Restoration of Bladder Function After Spinal Cord Injury: Simulation-Based Modeling and Interactive Programming Integration for Bladder Home-Training
Brief Title: SPARC Bladder Mapping and Training Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Susan Harkema PhD, Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17.1024; 1UH3NS116238-01 (NIH); 3OT2OD024898-01S5 (NIH); 1R01HL150581-01A1 (NIH)
Record Dates: First submitted 2018-02-25; First posted 2018-03-02 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injuries
Keywords: Epidural Stimulation; Bladder dysfunction; Spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Bladder Mapping and Training (Experimental): Individuals already implanted or newly implanted with a spinal cord epidural stimulator will receive epidural stimulation targeted at enhancing both the storage and voiding phase of micturition cycle.
  Interventions: Device: Epidural Stimulation

INTERVENTIONS:
Device: Epidural Stimulation — Spinal cord epidural stimulation will be administered through a multi-electrode array implanted in the epidural space over the dorsum of the spinal cord. An implanted package containing stimulating circuits, rechargeable battery, and wireless communication activates the electrodes (16 platinum electrodes arranged in three columns of [5-6-5]). The pattern of electrically active electrodes, as well as electrode voltage, stimulating frequency, and stimulating pulse width will be varied to facilitate effects toward bladder function.

SUMMARY:
The investigators propose to determine the electrode configurations that promote functional gains in the storage and voiding phases of lower urinary tract function as a result of activation of spinal circuits with spinal cord epidural stimulation in humans with spinal cord injury. The innovative approach and novel application of the Medtronic Specify 5-6-5 (16-electrode array) epidural device will allow the investigators to determine, with this early feasibility study, specific parameters of spinal cord epidural stimulation and approaches for bladder training needed for lower urinary tract function which will lay the groundwork for expedient translation of this promising technology to larger numbers of individuals with spinal cord injury who currently have limited treatment options. The current proposed study will increase the understanding of human lumbosacral spinal networks and guide the use of innovative therapeutic strategies that would be immediately available to not only improve the motor output during standing and walking but also ameliorate bladder dysfunction and thus improve quality of life in individuals after spinal cord injury.

DETAILED DESCRIPTION:
Deficits in urologic function after spinal cord injury impact quality of life and consistently ranks as a top priority issue in the spinal cord injury population. Bladder dysfunction may manifest as detrusor hyperreflexia (bladder contractions at low volumes, causing incontinence and smooth muscle hypertrophy), detrusor-sphincter dyssynergia (uncoordinated bladder and external urethral sphincter contractions, causing inefficient emptying and smooth muscle hypertrophy), decreased compliance (unable to store urine under appropriately low pressures) and loss of continence, requiring lifelong management, maintenance, and health care visits. Current therapeutic approaches aim to manage both the storage and voiding phases of bladder function and include intermittent catheterization, pharmacologic and surgical interventions. While most of these strategies are necessary for urological maintenance post-injury they oftentimes are associated with side effects and therefore remain inadequate. Therapies addressing recovery of function are still needed. The use of spinal cord epidural stimulation is a promising alternative approach to addressing the primary phases of bladder dysfunction. Additionally, the effects of spinal cord epidural stimulation on bladder alone is not known as its use has been directed towards the locomotor system. Thus, the overall objective of this study is to perform functional mapping in order to identify the spinal cord epidural stimulation configurations (anode/cathode selection, amplitude, frequency and pulse width) at the lumbosacral level that can promote neural control of bladder storage (capacity) and bladder emptying (voiding efficiency) after spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* stable medical condition without cardiopulmonary disease or dysautonomia that would contraindicate bladder training;
* clear indications that the period of spinal shock is concluded determined by presence of muscle tone, deep tendon reflexes or muscle spasms and discharged from standard inpatient rehabilitation;
* non-progressive supra-sacral SCI (i.e., upper motor neuron re bladder circuitry);
* AIS classification A or B;
* at least 2 years post spinal cord injury.

Exclusion Criteria:

* Painful musculoskeletal dysfunction, unhealed fracture, contracture, pressure sore or urinary tract infection that might interfere with mapping/training;
* Clinically significant depression or ongoing drug abuse;
* Pregnant at the time of enrollment or planning to become pregnant during the time course of the study
* Bladder Botox injections within the past year;
* Continent diversion procedures with or without bladder augmentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in bladder volume during filling cystometry at low filling pressures | 2 years
  The quantitative metric will be the percent changes in either residual volume (measured in ml) alone if no leak occurred or leak volume divided by leak plus residual volumes if a void occurred upon reaching capacity.

SECONDARY OUTCOMES:
Changes in Sexual Function | 2 years
  International SCI Data Set Questionnaire for Sexual Function
Changes in Bowel Function | 2 years
  International SCI Data Set Questionnaire for Bowel Function
Changes in Systolic Blood Pressure | 2 years
  Percent change without versus with epidural stimulation

OTHER OUTCOMES:
Changes in Renal Bladder Ultrasound | 2 years
  Measurements include kidney dimensions, parenchymal thickness, renal and aortic velocities, bladder size and thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Harkema, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/07/NCT03452007/ICF_002.pdf